CLINICAL TRIAL: NCT05910684
Title: Establishing Clinical Utility Evidence for Chronic Disease Management Testing: A CPV® and Chart Abstraction Randomized Controlled Trial
Brief Title: Establishing Clinical Utility Evidence for Chronic Disease Management Testing Patient Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00060013
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study will enroll primary care physicians practicing in the US from a population of participants who completed phase 1 of the study. All participants will keep their arm assignments from the phase 1 study. All eligible and consented participants will complete a round of three patient simulations.
  The intervention arm will have access to the Aegis test and will be asked to use this test on patients who meet the eligibility criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (No Intervention): These participants will complete their online simulations and treat their real-life patients without access to the Aegis test.
- Educational Materials and Test Access (Experimental): These participants will complete their online simulations and treat their real-life patients with access to educational materials and the Aegis test results. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Diagnostic Test: Aegis CDM Test and Educational Materials

INTERVENTIONS:
Diagnostic Test: Aegis CDM Test and Educational Materials — The Aegis CDM diagnostic test will be given to intervention participants to use on their patients. The participants will receive the results of the test through a web portal. Investigators will analyze the differences in quality of care between the control arm and the intervention arm.
  Arms: Educational Materials and Test Access

SUMMARY:
This is a national-level research study of primary care physicians. The purpose of this study is to assess the clinical evaluation and management (drug, procedures, counseling, and others) of a subset of common patient care indications.

DETAILED DESCRIPTION:
In the original study protocol (approved on October 19th, 2021), which the investigators are now referring to as Phase 1, the investigators measured changes in clinical practice using Clinical Performance and Value (CPVs) vignettes, described below. Phase 1 utilized simulated patients to determine clinical variation in the management of chronic cardiometabolic diseases and assessed the impact of the CDMT results on physicians' clinical decision-making.

CPVs are QURE's scientifically-validated measurement tool, first described in JAMA, 2000, and now used in scores of scientific investigations. In this research and derivative peer-reviewed publications, QURE's CPV studies efficiently measure clinical practice patterns among active physicians to determine if there is value in new technologies to payers.

This amendment allows us to ask the same physicians if they change their practice in an actual clinical setting.

Phase 2 extends the findings from Phase 1 by measuring the change in clinical practice using CPVs and securing data on practice patterns from abstracted medical records. the investigators will look for the same changes the investigators found in Phase 1 to determine the impact of CDMT on real-world clinical decisions and patient outcomes. The advantage of Phase 2 is that it leverages the same sample frame and the randomization by returning to the physicians in Round 1 who indicated that CDMT would change their practice. These physicians will be given, free of charge, the option of using CDMT on their real patients who share similar medical diagnoses as the CPV simulated patients. Phase 2 will thus provide patient-level data on the impact of medication adherence assessment on quality outcomes including, but not limited to, blood pressure control, blood sugar control, and parameters of disease progression

ELIGIBILITY:
Inclusion Criteria:

* Board-certified physician currently practicing in either Family Medicine or Internal Medicine.
* Have practiced as a board-certified physician in internal or family medicine or greater than 2 but less than 30 years
* Community/non-academic based practice setting
* ≥ 40 patients under care weekly
* Commonly treats patients with atrial fibrillation, coronary artery disease, congestive heart failure, diabetes, hypertension, and hyperlipidemia
* Patient HIPAA Authorization form signed upon initial enrollment into the provider's practice
* Practicing in the U.S.
* English-speaking
* Access to the internet
* Informed and voluntarily consented to be in the study

Exclusion Criteria:

* Not a board-certified physician
* Not practicing in the United States
* Not informed and voluntarily consented to be in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Chart abstraction measured variation in quantity of care | [19 months]
  Measuring the difference in the quality of care between the control arm and the intervention arm as measured by the number of care decisions made in the second round of chart abstraction.
  These care decisions might include decisions such as avoidance of invasive diagnostic tests, reductions in unneeded specialist referrals, increased diagnosis and treatment of drug-drug interactions, or care decisions related to costs.
Chart abstraction measured variation in quality of care | [19 months]
  Measuring the difference in the quality of care between the control arm and the intervention arm as measured by the quality of care decisions made in the second round of chart abstraction.
  These care decisions might include decisions such as avoidance of invasive diagnostic tests, reductions in unneeded specialist referrals, increased diagnosis and treatment of drug-drug interactions, or care decisions related to costs.
Chart abstraction measured variation in clinical decisions | [19 months]
  Measuring the variation in amount of evidence based clinical decisions among practicing primary care physicians in the assessment, recognition, and adjustment of treatment due to medication non-adherence and DDIs in patients with chronic cardiometabolic diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David RE, Ferrara KG, Schrecker J, Paculdo D, Johnson S, Bentley-Lewis R, Heltsley R, Peabody JW. Impact of medication nonadherence and drug-drug interaction testing on the management of primary care patients with polypharmacy: a randomized controlled trial. BMC Med. 2024 Nov 18;22(1):540. doi: 10.1186/s12916-024-03757-6. PMID 39551766